CLINICAL TRIAL: NCT06979648
Title: Effectiveness of Qualia Magnesium+® Supplementation on RBC Magnesium Levels: A Randomized Double-Blind Parallel Trial
Brief Title: Effectiveness of Qualia Magnesium+® Supplementation on RBC Magnesium Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: QLS-011
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Magnesium Deficiency
Keywords: Magnesium supplementation; magnesium
MeSH Terms: conditions — Magnesium Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qualia Magnesium+® (Active Comparator): Qualia Magnesium+® Supplement
  Interventions: Dietary Supplement: Qualia Magnesium+®
- Placebo (Placebo Comparator): Rice Flour
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Qualia Magnesium+® — Qualia Magnesium+® manufactured by Qualia Life Sciences
  Arms: Qualia Magnesium+®
Dietary Supplement: Placebo — Rice Flour
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled parallel trial designed to evaluate the effectiveness of Qualia Magnesium+® supplementation on red blood cell (RBC) magnesium levels in adults aged 21 and older. Approximately 100 participants with baseline RBC magnesium levels below 6.0 mg/dL will be randomly assigned to receive either Qualia Magnesium+ or a placebo. Participants will take 2 capsules daily in the evening, with or without food, for a duration of 12 weeks. The primary outcome is the between-group change in RBC magnesium levels from baseline to Week 12. Secondary outcomes include assessments of sleep quality, perceived stress, magnesium status, and safety and tolerability. Data collection will occur through lab bloodwork and electronic questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary, written, informed consent to participate in the study
* Agree to provide a valid cell phone number and are willing to receive communications through text
* Can read and write English
* Willing to complete questionnaires, records, and diaries associated with the study.
* Male and female participants aged 21 years and older
* Willing and able to visit a local blood draw facility for required blood sample collections
* Live within 20 miles of a suitable blood draw facility (such as Quest)
* RBC Magnesium levels below 6.0 mg/dL
* Willing to not consume any supplements containing magnesium starting about 2 weeks prior to the baseline magnesium blood test and continuing through the intervention period.
* Willing to not begin taking any new supplements during the study and continue taking any supplements they are currently using regularly with the exception of those containing magnesium

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
* Known food intolerances/allergy to any ingredients in the product
* Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, cancer
* Having had a significant cardiovascular event in the past 6 months
* Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines
* On immunosuppressive therapy
* Individuals who were deemed incompatible with the test protocol
* Adults lacking capacity to consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-21 (Estimated); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-09-21 (Estimated)

PRIMARY OUTCOMES:
Between-group change in RBC magnesium levels | 12 weeks
  To assess the between-group change in RBC magnesium levels from baseline to Week 12 following supplementation with Qualia Magnesium+ or placebo.

SECONDARY OUTCOMES:
To evaluate changes in sleep quality using the PROMIS Sleep Disturbance Short Form | 4, 8, and 12 weeks
To assess perceived stress levels with the PSS-10 | 4, 8, and 12 weeks
To evaluate changes in the magnesium status using the Magnesium Status Questionnaire | 4, 8, and 12 weeks
Side effect profile as measured by a custom Safety and Tolerability survey | 4, 8, and 12 weeks
  Number of participants with treatment-related adverse events as assessed by a score of 3 or greater on the Safety and Tolerability survey
To assess changes in serum magnesium levels | 4, 8, and 12 weeks
Between-group change in RBC magnesium levels | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Qualia Life Sciences, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No